CLINICAL TRIAL: NCT00976898
Title: Phase II Study of Proton Beam Irradiation for the Treatment of Unresectable Hepatocellular Cancer and Cholangiocarcinoma
Brief Title: Proton Beam Irradiation for the Treatment of Unresectable Hepatocellular Cancer and Cholangiocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); National Cancer Institute (NCI) (NIH); M.D. Anderson Cancer Center (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Hannah Roberts, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-131; P01CA021239 (NIH)
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Liver Cancer
Keywords: proton beam radiation
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Beam Irradiation (Experimental): This is a single arm study. All study participants will receive proton radiation therapy.
  Interventions: Radiation: Proton Beam Irradiation

INTERVENTIONS:
Radiation: Proton Beam Irradiation — Given once a day, 5 days a week, for 3 weeks

SUMMARY:
In this study the investigators will be studying the effects of proton beam radiation therapy. This is a very accurate kind of treatment that has been shown to affect less normal tissue than a photon radiation beam. The accuracy allows the investigators to more safely increase the amount of radiation delivered to eliminate cancer. This accuracy will potentially reduce side effects that participants would normally experience using photon radiation therapy. The purpose of this study is to determine if radiation using proton beam therapy will kill the cancer cells in the participants liver.

DETAILED DESCRIPTION:
* Participants will receive treatment as an outpatient in the Francis H. Burr Proton Center at the Massachusetts General Hospital, the MD Anderson Proton Therapy Center or the Roberts Proton Therapy Center at the University of Pennsylvania.
* Not everyone who participates in this study will be receiving the same dose of radiation. The dose received will be determined by the location of the tumor(s) within the liver.
* Proton Beam radiation therapy to the liver will be given once a day, 5 days a week (Monday-Friday), for 2 weeks.
* The following procedures will be performed once a week during treatment on days 1, 8 and 15, as well as on the last day of radiation: physical examination and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven unresectable or locally recurrent hepatocellular cancer or intrahepatic cholangiocarcinoma. Patients with a single lesion must be 12cm or less in greatest dimension. For patients with two lesions, no lesion may be greater than 10cm in greatest dimension. For patients with three lesions, no lesion may be greater than 6cm in greatest dimension. Patients may have single or multinodular tumors (up to 3). There must be no evidence of extrahepatic tumor. Portal vein involvement or thrombosis is allowed.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 20mm or greater with conventional techniques or as 10mm or greater with spiral CT scan.
* Patients may have had prior chemotherapy, targeted biological therapy, surgery, transarterial chemoembolization (TACE), radiofrequency ablation, or cryosurgery for their disease as long as it is greater than 4 weeks from first protocol radiation treatment (6 weeks for nitrosoureas or mitomycin C). Patients may not have had prior radiation to the affected area.
* 18 years of age or older
* Expected survival must be greater than three months
* ECOG Performance Status of 0, 1 or 2
* Normal organ and marrow function as outlined in the protocol
* If patient has underlying cirrhosis, only Child-Pugh classification Group A or Group B patients should be included in this study.
* Patients must be either surgically sterile or post-menopausal. Male and female patients of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of the study participation.
* Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin

Exclusion Criteria:

* Women who are pregnant or lactating
* Patients with evidence of non-hepatic metastatic disease
* Local conditions or systemic illnesses which would reduce the local tolerance to radiation treatment, such as serious local injuries, active collagen vascular disease, etc.
* Prior liver directed radiation treatment
* Patients may have no serious medical illness, which may limit survival to less than 3 months
* Patients may have no serious psychiatric illness/social situations which would limit compliance with study requirements
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other study agents
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-08; Primary Completion 2017-03 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah J. Roberts, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pennsylvania, Roberts Proton Facility, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Beam Irradiation
Started | 83
Completed | 78
Not Completed | 5
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Liver Transplant | 1
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Proton Beam Irradiation
Number analyzed (Participants) | 83
Age, Continuous [Median (Full Range); unit: years] | 67.6 [29.9 to 89.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 76
  Black | 4
  Asian | 1
  Hispanic (white or black) | 1
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 83
Underlying Liver Disease [Count of Participants; unit: Participants]
  Hepatitis C Virus (HCV) (± Others) | 28
  No HCV but Hepatitis B Virus (HBV) (± Others) | 6
  No HCV/HBV but Ethyl Hepatocellularalcohol (EtOH) | 8
  No HCV/HBV/EtOH but nonalcoholic steatohepatitis | 3
  Other | 2
  None | 36
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) score:
  * 0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  * 1 - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  * 2 - Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  Participants
    0 | 28
    1 | 52
    2 | 3
Child-Turcotte-Pugh Class [Count of Participants; unit: Participants] — Child-Turcotte-Pugh Class is used to evaluate the prognosis of chronic liver disease (primarily cirrhosis). Classes are determined using 5 clinical measures of liver disease with 1 to 3 points given for each measure, with more points given for less favorable clinical criteria. The 5 measures are total bilirubin, serum albumin, prothrombin time/international normalized ratio (INR), Ascites, and hepatic encephalopathy grade. The classes are A (5-6 points), B (7-9 points), and C (10-15 points) with 'A' having the best survival outcomes and C having the worst.
  Participants
    A | 66
    B | 15
    C | 0
    No Cirrhosis | 4
Disease Status [Count of Participants; unit: Participants]
  Locally Recurrent | 5
  Newly Diagnosed | 78
Number of Nodular Tumors [Count of Participants; unit: Participants]
  1 | 66
  2 | 15
  3 | 4
Previous Therapy [Count of Participants; unit: Participants]
  Any surgical resection | 4
  Any transarterial chemoembolization | 5
  Any radiofrequency ablation | 2
  Any chemotherapy | 27
  Any other | 15
  None | 45

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Local Control Rate
Description: The percentage of participants with local control after two years as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.0. The duration of control was measured from the start of treatment. Local control is the absence of local failure. Local Failure is defined as evidence of tumor growth/regrowth in any direction beyond that present of the pre-treatment imaging studies in the treated lesion(s).
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Beam Irradiation
Number analyzed (Participants) | 83
percentage of participants | 94.4 [87.2 to 98.2]

2. Primary Outcome: Median Overall Survival
Description: The median survival time in months as measured from the start of treatment until death due to any cause or until the participants is censored. Participants are censored at the date of their last follow-up.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Proton Beam Irradiation
Number analyzed (Participants) | 83
Months | 49.9 [17.8 to NA] — Upper bound not reached because of living subjects

3. Secondary Outcome: Number of Participants With Treatment Related Adverse Events ≥ Grade 3
Description: Summary of the proton radiation related grade 3 or greater adverse events that participants experienced. Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE v3).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Beam Irradiation
Number analyzed (Participants) | 83
Participants
  Liver Failure | 1
  Platelets | 1
  Ascites (nonmalignant) | 1
  Ulcer, GI - stomach | 1
  Bilirubin (hyperbilirubinemia) | 1

4. Secondary Outcome: Patterns of Failure
Description: A summary of the patterns of treatment failure, shown as the number of participants that fall into each category at the end of study follow-up
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Beam Irradiation
Number analyzed (Participants) | 83
Participants
  Alive, no progression | 26
  Distant metastases | 38
  Local failure and distant metastases | 3
  Isolated local failure | 5
  Dead of disease, no progression | 2
  Dead of other causes, no progression | 9

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from the start of treatment until 30 days after the last study visit. Radiation was delivered in 15 fractions Monday through Friday over a period of three weeks. Follow-up visits occurred at 1, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 months post treatment. Median follow-up was 19.5 months.
Description: Adverse events were assessed with the use of regularly scheduled visits which involved physical exams, CT and/or MRI scans, laboratory tests, and patient self reporting. If an adverse event did not match any of the existing CTCAE 3 terms, it was noted as being 'other'. Adverse events noted as being 'other' were only grouped together by organ system due to incomplete data about what specific adverse event was being recorded as 'other'.
Arm/Group | Proton Beam Irradiation
All-Cause Mortality (participants affected / at risk) | 11/83
Serious Adverse Events (participants affected / at risk) | 8/83
Other Adverse Events (participants affected / at risk) | 81/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Beam Irradiation (N=83)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Infection with unknown ANC - Abdomen NOS (Infections and infestations) | 1 (1)
Platelets (Investigations) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Beam Irradiation (N=83)
Alkaline phosphatase (Investigations) | 13 (40)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 11 (41)
Anorexia (Metabolism and nutrition disorders) | 38 (92)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 5 (10)
Ascites (non-malignant) (Gastrointestinal disorders) | 20 (43)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 21 (75)
Bilirubin (hyperbilirubinemia) (Investigations) | 18 (79)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 16 (47)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 8 (23)
Cardiac General - Other (Cardiac disorders) | 5 (14)
Constipation (Gastrointestinal disorders) | 14 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (23)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 13 (41)
Diarrhea (Gastrointestinal disorders) | 18 (31)
Distension/bloating, abdominal (Gastrointestinal disorders) | 16 (29)
Dizziness (Nervous system disorders) | 11 (25)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 23 (38)
Edema: limb (General disorders) | 22 (60)
Encephalopathy (Nervous system disorders) | 5 (6)
Extremity-lower (gait/walking) (General disorders) | 5 (12)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 67 (316)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 9 (25)
Fracture (Injury, poisoning and procedural complications) | 7 (20)
Gastrointestinal - Other (Gastrointestinal disorders) | 13 (29)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 (34)
Heartburn/dyspepsia (Gastrointestinal disorders) | 11 (25)
Hemoglobin (Blood and lymphatic system disorders) | 9 (25)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 13 (32)
Hypertension (Vascular disorders) | 5 (10)
Hypotension (Vascular disorders) | 9 (16)
Insomnia (Psychiatric disorders) | 10 (25)
Leukocytes (total WBC) (Investigations) | 7 (21)
Memory impairment (Nervous system disorders) | 5 (9)
Metabolic/Laboratory - Other (Investigations) | 5 (10)
Mood alteration - Anxiety (Psychiatric disorders) | 10 (22)
Depression (Psychiatric disorders) | 8 (24)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 8 (13)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 7 (15)
Nausea (Gastrointestinal disorders) | 40 (104)
Neuropathy: sensory (Nervous system disorders) | 5 (18)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 (12)
Pain - Abdomen NOS (Musculoskeletal and connective tissue disorders) | 36 (136)
Pain - Back (Musculoskeletal and connective tissue disorders) | 12 (21)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 9 (17)
Pain - Chest/thorax NOS (General disorders) | 6 (8)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 9 (19)
Pain - Head/headache (Nervous system disorders) | 6 (11)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 8 (16)
Pain - Other (General disorders) | 14 (33)
Platelets (Investigations) | 24 (90)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 7 (13)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 (13)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 7 (17)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (8)
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 5 (5)
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 51 (194)
Rigors/chills (General disorders) | 9 (13)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8 (16)
Somnolence/depressed level of consciousness (Nervous system disorders) | 5 (5)
Ulceration (Skin and subcutaneous tissue disorders) | 5 (8)
Urinary frequency/urgency (Renal and urinary disorders) | 8 (18)
Urine color change (Renal and urinary disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 18 (22)
Weight loss (Investigations) | 12 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT00976898/Prot_SAP_000.pdf